CLINICAL TRIAL: NCT03718507
Title: A Single-centre, Randomized Pilot Study on the Effects of Different Premedication Treatments for Less Invasive Surfactant Administration (LISA) on Pain, Cerebral Tissue Oxygenation and Cortisol Levels in Preterm Infants
Brief Title: Study on the Effects of Different Premedication for LISA on Stress and Cerebral Tissue Oxygenation in Preterm Infants
Acronym: SAFE LISA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no recrutiment started
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Dr. Ilia Bresesti, Dr, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SL2018PS
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Distress Syndrome; Surfactant Deficiency Syndrome Neonatal; Near Infrared Spectroscopy
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Atelectasis | interventions — Fentanyl; Atropine; Sucrose; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP Fentanyl (Active Comparator): patients will receive atropine (0.01-0.02 mg/kg i.v. bolus) and fentanyl (0.5-2 mcg/kg i.v. in 5 minutes) before LISA in addition to standard care (wrapping). NIRS will be monitored during the whole procedure, which will be video-recorded.
  Interventions: Drug: Fentanyl
- GROUP Sucrose (Experimental): patients will be given atropine (0.01-0.02 mg/kg i.v. bolus) and oral sucrose 24% (0.5 ml) 2 minutes before LISA in addition to standard care (wrapping). NIRS will be monitored during the whole procedure, which will be video-recorded.
  Interventions: Drug: Sucrose 24% Oral Solution

INTERVENTIONS:
Drug: Fentanyl — atropine (0.01-0.02 mg/kg i.v. bolus) and fentanyl (0.5-2 mcg/kg i.v. in 5 minutes)
  Other Names: atropine
  Arms: GROUP Fentanyl
Drug: Sucrose 24% Oral Solution — 0.5 ml given orally 2 minutes before LISA procedure
  Other Names: atropine
  Arms: GROUP Sucrose

SUMMARY:
Given the popularity that LISA technique has gainig in worldwide neonatal units, the lack of evidence regarding its premedication is becoming even more relevant to provide the best care to premature infants.

Objective of this clinical trial is to establish the best premedication for LISA procedure considering neonatal pain assessed with premature infants pain scale, salivary cortisol levels as an indicator of stress and crSO2 values as indicators of cerebral oxygenation. Moreover, we aim to verify if sucrose 24% given orally is an effective tool for pain management in preterm neonates also in more invasive procedure, comparable to pharmacological treatment.

DETAILED DESCRIPTION:
In the last decades, one of the most relevant interventions which have led to a significant increase in preterm infants survival rate is the introduction of surfactant replacement therapy.

Nowadays, given the trend towards the less invasive respiratory support also for low and extremely low gestational age infants, the use of intubation and prolonged mechanical ventilation has been minimized. In fact, bronchopulmonary dysplasia (BPD) has been proved to be closely related to prolonged intubation and it is one of the main problem clinicians must face with. This is the reason why the INSURE technique was introduced as a routine care procedure in neonatal units. In fact, INSURE is the acronym for INtubation - SURfactant administration-Extubation. This technique ensures the baby the positive effects of surfactant on respiratory mechanics minimizing the intubation length. However, the INSURE procedure still involves intubation, meaning that it is still invansive and some infants cannot be extubated immediately afterward. Thus, lately new technique for surfactant administration has been introduced. The most extensively studied are the so-called less invasive surfactant administration (LISA) and minimally invasive surfactant therapy (MIST). With these procedures, infants receive non-invasive continuous positive airway pressure (CPAP) treatment, while being given intratracheal surfactant via a feeding tube or small catheter. Although the paucity of literature available to date, for extremely preterm infants LISA has shown to be able to reduce the need for intubation, ventilation and supplemental oxygen when compared with the standard technique of rescue intubation and ventilation. In comparison with the INSURE procedure the less invasive surfactant administration was associated with a reduced need for ventilation and reduced risk of BPD.

Even if this technique can provide the gentlest treatment presently available in administering surfactant, it implies laryngoscopy and somewhat discomfort. The importance of proper care in managing preterm infants, especially during painful procedures, has been well demonstrated and all the caregivers have to be even more committed to this aspect.

Pain in neonates is usually assessed through pain scales and using clinical parameters such as pulse oximetry (SatO2) and Heart Rate (HR). Since pain scores are subject to caregivers' individual perception and parameters can be influenced by other clinical underlying condition, especially in preterm infants, determination of cortisol concentration could be a useful alternative.

Cortisol is the major glucocorticoid produced in the adrenal cortex. Cortisol production has a circadian rhythm, with levels peaking in the early morning and dropping to lowest values at night. Levels rise independently of circadian rhythm in response to stress.

There is convincing evidence that providing neonates with oral glucose during painful procedure reduces the stress related to the procedure itself, without serious side effects or harms related to this intervention. Different concentrations of glucose solution are currently available and have been used in neonatal field.

To date, there is still high debate on the need to provide sedation to babies undergoing LISA, and lack of evidence available regarding the optimal premedication. Some Authors report to use LISA technique without any sort of sedation, while others perform it with the same sedation they use for INSURE method.

Moreover, there is lack of evidence in regard to the effects of this method on cerebral oxygenation, which can be easily monitored using NIRS (near infrared spectroscopy).

Since LISA technique's popularity is increasing, we believe that there is urgent need to better clarify how this approach can be performed in the gentlest way.

Given these premises, we indeed speculate that oral glucose as a premedication for LISA procedure could be an intriguing alternative to standard sedation.

Objective of this clinical trial is to establish the best premedication for LISA procedure considering neonatal pain assessed with premature infants pain scale, salivary cortisol levels as an indicator of stress and crSO2 values as indicators of cerebral oxygenation. Moreover, we aim to verify if sucrose 24% given orally is an effective tool for pain management in preterm neonates also in more invasive procedure, comparable to pharmacological treatment.

Evaluation of the efficacy of non-pharmacological sedation will lead to:

* a gentler approach for preterm babies and a better understanding of LISA technique
* an improvement in pain management, where sucrose can be applied for several painful procedures of different degrees of invasiveness, not only in the mildest ones
* a significant reduction in prolonged ventilation due to surfactant administration's pharmacological sedation
* a safer use of surfactant administration also in level II neonatal unit, since the risk for subsequent need of invasive respiratory support due to excessive sedation would be considerably reduced
* a significant economic impact on public health care system, for the inferior cost of oral sucrose
* a relevant decrease of the onset and subsequent public cost of BPD, if data about LISA technique capability to reduce it will be further confirmed.
* Primary Outcome:

Verify which is the best premedication for LISA procedure to reduce neonatal pain.

* Secondary Outcomes:
* Verify the effects of different forms of premedication on cerebral oxygenation during LISA procedure
* Verify the effects of different forms of premedication on cortisol levels before and after LISA procedure
* Verify the efficacy of sucrose 24% in pain control during more invasive procedures
* Verify the influence of premedication on adverse events' occurrence during LISA procedure
* Verify the effects of different pre-medications on the ease in administering surfactant with LISA technique (time required, number of attempts, …)

Trial Design:

An investigator-initiated randomized, single center, pilot study that will enroll 20 preterm neonates between 27 and 29+6 weeks of gestation.

Multiple births will be randomised into the same treatment arm.

Trial Interventions:

* Study group 1: patients will receive atropine (0.01-0.02 mg/kg i.v. bolus) and fentanyl (0.5-2 mcg/kg i.v. in 5 minutes) before LISA in addition to standard care (wrapping). NIRS will be monitored during the whole procedure
* Study group 2: patients will be given atropine (0.01-0.02 mg/kg i.v. bolus) and oral sucrose 24% (0.5 ml) 2 minutes before LISA in addition to standard care (wrapping). NIRS will be monitored during the whole procedure.

All the procedure will be videorecorded and subsequently analyzed

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonate 27-29+6 weeks AND
* Need for non-invasive respiratory support (CPAP or nHFT) AND
* Need for surfactant according to the unit guidelines AND
* Written informed consent

Exclusion Criteria:

* No written informed consent and/or
* Severe malformation of the upper/lower airways, brain and/or heart and/or lung and/or prenatal cerebral injury.

Ages: 27 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-02-20 (Estimated)

PRIMARY OUTCOMES:
PIPP SCALE score | during the LISA procedure
  Verify which is the best premedication for LISA procedure to reduce neonatal pain.

IPD SHARING:
Plan to Share IPD: No